CLINICAL TRIAL: NCT02728960
Title: TBI Biological Diagnosis Via High Definition Tractography Asymmetry Screening
Brief Title: Traumatic Brain Injury Biological Diagnosis Via High Definition Tractography Asymmetry Screening
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study under review. Temporarily suspended
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 12-03539
Record Dates: First submitted 2016-03-08; First posted 2016-04-06 (Estimated); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Traumatic Brain Injury (Experimental): Documented history of Traumatic Brain Injury
  Interventions: Procedure: MRI of the Brain (No Contrast) Scan
- Normal Controls (Active Comparator): No prior history of concussion, TBI, blast exposure, stroke, or other major neurological disorder
  Interventions: Procedure: MRI of the Brain (No Contrast) Scan
- Sequence Development Volunteers (Active Comparator)
  Interventions: Procedure: MRI of the Brain (No Contrast) Scan

INTERVENTIONS:
Procedure: MRI of the Brain (No Contrast) Scan — DSI data will be acquired on 3T Tim Trio System (Siemens) using a 32-channel coil

SUMMARY:
The primary purpose of this study is to validate the High Definition Fiber Tracking (HDFT/HDFTAS) technology, so that faster, more reliable diagnosis can be implemented in Traumatic Brain Injury (TBI). This study will involve Traumatic Brain Injury Patients and normal controls, in addition to 30 pilot participants who will be undergoing MRI in order to develop a statistically sound range for the metrics derived from HDFT.

DETAILED DESCRIPTION:
This descriptive study sponsored by the United States Department of Defense involves the examination of TBI participants and normal control participants through MRI (Without Contrast) scanning. Normal controls are essential to develop a statistically sound range for the metrics derived from High Definition Fiber Tracking (HDFT). TBI subjects will undergo 1 MRI scan and normal controls will be asked to undergo 1 MRI scan. The study will involve blinded evaluations of results to determine the ability of HDFT imaging methods to evaluate TBI.

In addition to the TBI and normal controls evaluated in this research study, investigators will be running 30 pilot participants. These participants will be undergoing MRI in order to streamline our pulse sequence and calibrate the MRIs. This is part of the technical development for the project and will occur before the recruitment of TBI subjects and normal controls for comparison. Data from the pilot subjects will not serve as control data for the TBI subjects.

ELIGIBILITY:
Inclusion Criteria TBI subjects:

* Documented history of TBI (for Chronic).
* No MRI contraindications such as implanted ferrous metal, pacemakers, body weight above 125 Kg, (might not fit in the scanner), or concerns about claustrophobia.

Exclusion Criteria TBI subjects:

* Inability or unwillingness of subject to provide written informed consent.
* History of penetrating gunshot wound.

Inclusion Criteria Control subjects:

* No prior history of concussion, TBI, blast exposure, stroke, or other major neurological disorder.
* No MRI contraindications such as implanted ferrous metal, pacemakers, body weight above 125 Kg, (might not fit in the scanner), or concerns about claustrophobia.

Exclusion Criteria TBI subjects:

* Inability or unwillingness of subject to provide written informed consent.
* History of concussions, stroke, or penetrating gunshot wound.

Inclusion Criteria Sequence Development Subjects:

* No MRI contraindications such as implanted ferrous metal, pacemakers, body weight above 125 Kg, (might not fit in the scanner), or concerns about claustrophobia.

Exclusion Criteria Sequence Development Subjects:

* Inability or unwillingness of subject to provide written informed consent
* Contra-indication to MR imaging, such as ferrous metal, pacemakers, body weight above 125 Kg or concerns

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Diagnosis reliability measured by MRI scanning data results | 2 Hours
Amount of white matter damage using HDTAS DSI diffusion evaluation of volume and connectivity across 40 fiber tracts over 150 brain regions. | 2 Hours
  Tract anomalies will be coded as significant differences either to normative data of the tract or expected left/right ratio of tract axonal volume. White matter damage will first be quantified through HDFT evaluation of volume and connectivity across 40 fiber tracts over 150 brain regions
Comparison of severity of subjects with TBI using Diffusion Tension Imaging (DTI) | 2 Hours

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Boada, PhD, Principal Investigator — New York University Medical School